CLINICAL TRIAL: NCT06602700
Title: Effects of High-intensity Interval Training and Moderate-intensity Continuous Training on Functioning of Attentional Networks and Heart Rate Variability in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2023067H
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Adults
Keywords: high-intensity interval training; moderate-intensity continuous training; attention networks; heart rate variability

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HIIT intervention (Experimental)
  Interventions: Behavioral: HIIT
- MICT intervention (Experimental)
  Interventions: Behavioral: MICT
- Rest control (No Intervention)

INTERVENTIONS:
Behavioral: HIIT — high-intensity interval training
  Arms: HIIT intervention
Behavioral: MICT — moderate-intensity continuous training
  Arms: MICT intervention

SUMMARY:
This study investigated the effects of HIIT and MICT on functioning of attentional networks and explored the relationship between heart rate variability (HRV) and these networks in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected-to-normal vision
* normal auditory function without any reading disorders
* right-handed

Exclusion Criteria:

* color blindness
* color weakness
* dyslexia
* history of smoking
* cardiovascular diseases
* personal or family history of mental illness

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
reaction times of the ANT-I task | immediately after interventions
  ANT-I: Attention Network Test for Interactions
accuracy of the ANT-I task | immediately after interventions
  ANT-I: Attention Network Test for Interactions
HR | immediately after interventions
  HR: heart rate
heart rate variability | immediately after interventions

CONTACTS AND LOCATIONS:
Locations (1):
- Sports, Exercise and Brain Sciences Laboratory, Sports Coaching College, Beijing Sport University, Beijing 100084, China, Beijing, Haidian District, China